CLINICAL TRIAL: NCT04211519
Title: Mersin University Clinical Research Ethics Committee
Brief Title: Analysis of Bacterial Microbiome of Endodontically Infected Primary and Permanent Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Ebru Delikan, Ebru Delikan, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017/234
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Endodontic Disease; Endodontic Inflammation
Keywords: Endodontic disease; Microbiome; Permanent teeth; Primary teeth
MeSH Terms: conditions — Dental Pulp Diseases; Pulpitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Permanent teeth group (Experimental): For the disinfection of teeth, 30% hydrogen peroxide and 2.5% sodium hypochlorite solution were used for 30 seconds each. Then, 5% sodium thiosulfate solution was used to inactivate the disinfectant agents. Cavity preparation and root canal access were accomplished using sterile high-speed diamond burs under water cooling. Microbial samples were taken immediately by the same researcher from the largest root canal under strict aseptic conditions by using paper point method. Sterilized minimum four paper points were placed to the same level in root canal and the root canal content was absorbed. Each paper point was kept into the canal for at least 30 seconds. Then, paper points were placed into the Eppendorf tubes and refrigerated at -80 °C within 10 min.
  Interventions: Diagnostic Test: sampling
- Primary teeth group (Experimental): For the disinfection of teeth, 30% hydrogen peroxide and 2.5% sodium hypochlorite solution were used for 30 seconds each. Then, 5% sodium thiosulfate solution was used to inactivate the disinfectant agents. Cavity preparation and root canal access were accomplished using sterile high-speed diamond burs under water cooling. Microbial samples were taken immediately by the same researcher from the largest root canal under strict aseptic conditions by using paper point method. Sterilized minimum four paper points were placed to the same level in root canal and the root canal content was absorbed. Each paper point was kept into the canal for at least 30 seconds. Then, paper points were placed into the Eppendorf tubes and refrigerated at -80 °C within 10 min.
  Interventions: Diagnostic Test: sampling

INTERVENTIONS:
Diagnostic Test: sampling — sampling from endodontically infected primary and permanent teeth by using paper point method

SUMMARY:
Recognition of community profiles in endodontic infections may allow a better understanding of the pathogenesis of the disease and the establishment of more effective treatment protocols.

Therefore, the aim of the present study was to investigate bacterial diversity in endodontically infected primary and permanent teeth using 16S rRNA gene sequencing and QIIME 2TM (Quantitative Insights Into Microbial Ecology 2) bioinformatics pipeline

DETAILED DESCRIPTION:
Endodontic infections are defined as an infection of the pulp and periapical tissues. This infection is caused by microorganisms that invade the pulp via dental caries or dental trauma. In these mixed population infections, anaerobic bacteria have been reported to be conspicuously dominant and the number of microorganisms per canal may vary. Traditionally, the endodontic microbiome has been identified by culture-based (phenotype-based) techniques. Inability to cultivate approximately 40-55% of bacteria in the endodontic microbiome, bias or inexperience of researchers may limit the results of cultural research. Microbiome-based new generation sequencing (NGS), which was initially used in ecological studies, has been widely used in recent years to identify bacterial diversity using the 16S ribosomal RNA (rRNA) gene in endodontic infections microbiome, bias or inexperience of researchers may limit the results of cultural research. There are few studies investigating the endodontic microbiome in primary teeth. However, to the best of our knowledge, to date, there is no metagenomic study that investigates the endodontic microbiome of the primary and permanent teeth. It is a still question of whether there is a difference in the endodontic microbiomes during the mixed dentition period when both dentition types can be seen.

ELIGIBILITY:
Inclusion Criteria:

* have intact roots or <1/3 of physiological root resorption
* have clinical crowns that permit effective rubber dam isolation
* no mobility, fistula, pus discharge, gingival swelling, periapical abscess or internal resorption.

Exclusion Criteria:

* have marginal periodontitis, a history of pharmacological treatment, antibiotics or fluoride intake within the last 2 months
* a history of cancer, diabetes or immunodeficiency disorders

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Comparison of microbiome composition of endodontically infected primary and permanent tooth canal | 6 months
  Analysis of the profile of microbial populations based on 16S rRNA gene analysis in endodontically infected permanent and primary teeth

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan Üniversitesi, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided